CLINICAL TRIAL: NCT07233655
Title: A Randomized, Double-blind, Placebo-controlled Phase IIa Study to Evaluate the Efficacy and Safety of SHR-3045 Injection in Patients With Moderate to Severe Active Rheumatoid Arthritis
Brief Title: A Phase II Trial of SHR-3045 Injection in Patients With Rheumatoid Arthritis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-3045-201
Record Dates: First submitted 2025-11-13; First posted 2025-11-18 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Moderate to Severe Active Rheumatoid Arthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-3045 Injection Group (Experimental): SHR-3045 injection in different doses.
  Interventions: Drug: SHR-3045 Injection
- SHR-3045 Injection Placebo Group (Placebo Comparator): SHR-3045 injection placebo in different doses.
  Interventions: Drug: SHR-3045 Injection Placebo

INTERVENTIONS:
Drug: SHR-3045 Injection — SHR-3045 injection.
  Arms: SHR-3045 Injection Group
Drug: SHR-3045 Injection Placebo — SHR-3045 injection placebo.
  Arms: SHR-3045 Injection Placebo Group

SUMMARY:
This study is ongoing to explore the efficacy and safety of different strengths of SHR-3045 injection in moderate to severe active rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form before the start of activities related to this study, be able to understand the procedures and methods of this study, and be willing to strictly follow the clinical research protocol to complete this study.
2. Age 18 to 75 years (including both ends) at the time of signing the informed consent form, with no gender restrictions.
3. Suffer from moderate to severe active rheumatoid arthritis (RA).
4. Have shown an inadequate response or intolerance to at least one conventional synthetic disease-modifying antirheumatic drug (csDMARD), biologic disease-modifying antirheumatic drug (bDMARD), or targeted synthetic disease-modifying antirheumatic drug (tsDMARD) during screening.
5. Have a body mass index (BMI = weight (kg) / height² (m²)) of ≥ 18 kg/m² at the time of screening.

Exclusion Criteria:

1. General conditions: (1) Pregnant or breastfeeding women; (2) Have not used or refused to use the contraceptive measures specified in the study protocol within 6 months after the last intake of medication (except for subjects or partners who are infertile); (3) Drug abuse; (4) The researcher judges that there are factors affecting the safety and efficacy evaluation of the study drug.
2. Within 4 weeks prior to the random visit, the following conditions are identified in laboratory tests and 12-lead electrocardiogram (ECG): (1) White blood cell count < 3.0 × 10⁹/L; (2) Neutrophil count < 1.5 × 10⁹/L; (3) Hemoglobin < 90.0 g/L; (4) Platelet count < 100 × 10⁹/L; (5) Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 times the upper limit of normal (ULN), or total bilirubin (T-BIL) > 1.5 times the upper limit of normal (ULN); (6) Estimated glomerular filtration rate (eGFR) calculated by the Modification of Diet in Renal Disease (MDRD) formula < 60 mL/min/1.73 m² (see details in Section 13.4 of the Appendix); (7) Glycated hemoglobin (HbA1c) ≥ 8.0%; (8) Positive anti-hepatitis C virus (HCV) antibody with HCV RNA exceeding the upper limit of normal, positive human immunodeficiency virus (HIV) antibody, or positive syphilis antibody; (9) 12-lead ECG indicates clinically significant abnormalities that may affect the safety of the subject, including but not limited to acute myocardial ischemia, myocardial infarction, severe arrhythmia, or significant QTc prolongation (QTc > 500 ms).
3. Any of the following medical histories or concurrent diseases exist: (1) Allergy to the study drug or any of its components; (2) Other systemic inflammatory diseases or autoimmune diseases except rheumatoid arthritis (RA); (3) Tuberculosis (TB) or latent tuberculosis infection; (4) History of non-tuberculous mycobacterial infection or opportunistic pathogen infection within 6 months before screening; (5) History of recurrent herpes zoster, disseminated herpes zoster or disseminated herpes simplex; (6) History of potential or active granulomatous inflammation, such as histoplasmosis, coccidioidomycosis, etc.; (7) History of chronic infection requiring treatment within 12 months before screening; (8) History of infection (viral, bacterial, fungal, parasitic) within 3 months before randomization, with hospitalization and/or parenteral systemic antimicrobial treatment; history of systemic antimicrobial treatment within 2 weeks before randomization; or open drainage wounds or ulcers at screening; or presence of joint prosthesis infection; (9) History of lymphoproliferative disorders; (10) History of malignant tumors or cancer; (11) Severe gastrointestinal diseases, or previous treatments that may affect drug absorption, history of gastrointestinal bleeding; (12) Moderate to severe congestive heart failure; (13) Uncontrolled grade 2 or higher hypertension; (14) History of thrombotic diseases within 12 months before randomization; (15) Cardiovascular or cerebrovascular events leading to hospitalization within 12 months before randomization; (16) History of organ transplantation; (17) Major surgery within 3 months before randomization, or planned major surgery during the study period; (18) Severe mental or neurological disorders or diseases (including alcoholism), unwillingness to communicate or language barriers, inability to fully understand and cooperate.
4. The use of any of the following drugs or participation in clinical research (defined as signing the informed consent form): (1) Use of cytotoxic drugs; (2) Use of etanercept or etanercept biosimilar within 4 weeks before randomization; use of infliximab or infliximab biosimilar, adalimumab or adalimumab biosimilar, golimumab, certolizumab, tocilizumab, sarilumab, or abatacept within 8 weeks before randomization; use of rituximab within 1 year before randomization; (3) Use of other drugs known to have strong immunosuppressive or immunomodulatory effects within 3 months before randomization, except for the above-mentioned drugs; (4) BCG vaccination within 12 months before screening; exposure to other live vaccines or attenuated live vaccines within 3 months before randomization; or plan to receive live vaccines or attenuated live vaccines during the study period; (5) Participation in any other drug or medical device clinical research within 3 months before randomization or within 5 half-lives of the drug (whichever is longer); (6) Intramuscular or intravenous administration of glucocorticoids within 4 weeks before randomization; (7) Intra-articular injection treatment (such as glucocorticoids, hyaluronic acid, etc.) within 4 weeks before randomization; (8) Use of traditional Chinese medicine preparations for the treatment of RA (such as Tripterygium wilfordii, total glucosides of paeony, sinomenine, etc.) or traditional Chinese medicine or Chinese patent medicine within 4 weeks before randomization; (9) Systemic interferon treatment within 4 weeks before randomization; (10) Use of strong opioids.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-19 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
The percentage of subjects who achieved a 20% improvement in the American College of Rheumatology Rheumatoid Arthritis (RA) disease activity assessment core set. | After 14 weeks of treatment.

SECONDARY OUTCOMES:
The percentage of subjects achieving a 20% improvement in the American College of Rheumatology (ACR) criteria for rheumatoid arthritis (RA) disease activity. | Within 169 days after administration.
The percentage of subjects achieving a 50% improvement in the American College of Rheumatology (ACR) criteria for rheumatoid arthritis (RA) disease activity. | Within 169 days after administration.
The percentage of subjects achieving a 70% improvement in the American College of Rheumatology (ACR) criteria for rheumatoid arthritis (RA) disease activity. | Within 169 days after administration.
Changes in the 28-joint disease activity score (DAS28) levels from the baseline. | Within 169 days after administration.
Changes in the C-reactive protein (CRP) levels from the baseline. | Within 169 days after administration.
Changes in the erythrocyte sedimentation rate (ESR) levels from the baseline. | Within 169 days after administration.
Changes in the simplified disease activity index (SDAI) score from the baseline. | Within 169 days after administration.
Changes in the clinical disease activity index (CDAI) score from the baseline. | Within 169 days after administration.
Adverse events (AEs). | Within 169 days after administration.
Blood drug concentration of SHR-3045. | Within 169 days after administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People 's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided